CLINICAL TRIAL: NCT03245021
Title: First-line Treatment for Grade 1-3A Follicular Lymphoma Using Opdivo (Nivolumab) Plus Rituximab: The 1st FLOR Study
Brief Title: Nivolumab Plus Rituximab in First-line Follicular Lymphoma gr 1-3A
Acronym: 1stFLOR
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Eliza Hawkes (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Dr. Eliza Hawkes, Chief Principal Investigator, Austin Health
Organization: Austin Health (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-676
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Nivolumab; Rituximab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label (Other): Opdivo - Single-arm open label study
  Interventions: Drug: Opdivo

INTERVENTIONS:
Drug: Opdivo — All patients will receive:
  Nivolumab 240mg IV q2-weekly for four cycles
  Patients in complete remission (CR):
  Nivolumab 240mg IV q2-weekly for four further cycles (8 in total)
  Patients with partial response (PR), stable disease (SD), asymptomatic or minor progressive disease (PD) post 4cycles receive:
  Nivolumab 240mg IV plus rituximab 375mg/m2 IV q2-weekly for four cycles
  Patients in CR:
  Nivolumab 240mg IV q2-weekly for four further cycles (8 in total)
  Patients with PR, SD, asymptomatic or minor PD post 4 cycles receive:
  Nivolumab 240mg IV plus rituximab 375mg/m2 IV q2-weekly for four cycles
  Other Names: Rituximab

SUMMARY:
Firstline treatment for grade 13a Follicular Lymphoma using Opdivo (nivolumab) plus Rituximab: The 1st FLOR trial

DETAILED DESCRIPTION:
This study will involve participants with a condition called Follicular NonHodgkin Lymphoma (Follicular Lymphoma).

The main purpose of this study is to see if it is safe to give drug Nivolumab before and in combination with drug Rituximab and to see how effective Nivolumab is in patients who have had no previous drug treatment for their lymphoma. In particular, we will be monitoring for any specific side effects which may be increased by adding Nivolumab to Rituximab treatment, including monitoring of the immune system.

Participants will be reviewed at baseline and prior to each cycle of treatment for toxicity, scans will be performed at baseline, after 4 cycles of nivolumab, after 8 cycles of nivolumab +/rituximab and at 6 months post induction treatment phase and following completion of treatment, participants will be followed up for a total of 5 years (every 3 months for 2 years, every 6 months for 3 years). In participants with relapsed disease, these will be followed for survival every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically proven Follicular non Hodgkin lymphoma (FL) grades 1-3A according to the current World Health Organization classification.29 The B cell nature of the proliferation must be verified by the positivity with an anti-CD20 antibody.
3. No previous chemotherapy, or other investigational drug for this indication apart from focal radiotherapy.
4. Stage II-IV disease (Ann Arbor criteria). Stage II disease must not be encompassable in a single radiotherapy field and being considered for definitive radiotherapy.
5. Eastern Collaborative Oncology Group (ECOG) performance status 0 to 1 unless attributable to lymphoma, in which case patients of performance status 2 are also eligible.
6. Deemed to need treatment by treating investigator. Reasons for treatment can include, but are not limited to:

a. Any nodal or extranodal tumour mass >7cm AND/OR multiple extranodal disease sites b. Involvement of at least 3 sites each with diameter >3cm c. Symptomatic splenic enlargement d. Organ involvement/compression e. Ascites or pleural effusion f. Lactate Dehydrogenase (LDH) elevated g. Presence of systemic symptoms h. Disease progression in preceding 3 months i. Evidence of marrow infiltration with marrow compromise. (eg Hb, WBC or plt count below lower limit of institutional normal range).

g) Adequate bone marrow function including:

1. Haemoglobin >9.0 g/dL
2. White blood cells (WBC) ≥2000/μL
3. Neutrophils >1.5 x 109/L
4. Platelets >100 x 109/L at the time of study entry, unless attributed to bone marrow infiltration by lymphoma.

h) Adequate renal function with serum creatinine ≤1.5 x ULN or creatinine clearance (CrCl) ≥ 40mL/min (using Cockroft-Gault formula) Female CrCl = (140 - age in years) x weight (kg) x 0.85 72 x serum creatinine (mg/dL) Male CrCl = (140 - age in years) x weight (kg) x 1.00 72 x serum creatinine (mg/dL) i) Adequate hepatic function with AST/ALT ≤3x ULN and total bilirubin ≤1.5 x ULN (except subjects with Gilbert syndrome, who can have a total bilirubin ≤3 mg/dL or ≤51.3 μmol/L) j) Life expectancy > 3 months. k) Patients of childbearing potential willing to adhere to contraceptive precautions

1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment
2. Women must not be breastfeeding
3. WOCBP must use appropriate method(s) of contraception to avoid pregnancy for 23 weeks (30 days plus five half-lives of nivolumab) post-treatment completion
4. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. They must agree to adhere to contraception for a period of 31 weeks after the last day of nivolumab.
5. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, they must still undergo pregnancy testing as described in this section.

l) Written, informed consent.

Exclusion Criteria:

1. Grade 3B follicular lymphoma, transformed follicular lymphoma, other indolent lymphomas.
2. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
3. Central nervous system, meningeal involvement or cord compression by lymphoma.
4. Patients with active, known or suspected autoimmune disease. Patients with well controlled type I diabetes mellitus, coeliac disease, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, vitiligo or psoriasis not requiring systemic treatment, or other conditions not expected to recur in the absence of an external trigger are permitted to enrol.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Past history of interstitial lung disease.
7. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
8. Any other serious active disease.
9. Any positive test result for hepatitis B or hepatitis C virus during screening indicating acute or chronic infection.
10. Any positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
11. Any history of severe hypersensitivity reactions to other monoclonal antibodies. A history of allergy or intolerance (unacceptable AEs) to study drug components or Polysorbate-80-containing infusions
12. Medical or psychiatric conditions that compromise the patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility and safety of combination nivolumab and rituximab as determined by the proportion of toxicity grade 3 or higher per CTCAE v4.0 occurring on induction treatment (ie first 16 weeks of therapy) | 1st 16 weeks of therapy
  As determined by rate of toxicity grade 3 or higher per CTCAE v4.0

SECONDARY OUTCOMES:
Overall toxicity | 5 years
  As determined by rate of toxicity grade 3 or higher per CTCAE v4.0
Response rate | 1st 16 weeks of therapy
  Response Rate to Nivolumab + Rituximab according to the Lugano classification for Response Criteria for Non-Hodgkin Lymphoma
Complete response rate | 6 months post completion of induction treatment
  Response Rate to Nivolumab + Rituximab according to the Lugano classification for Response Criteria for Non-Hodgkin Lymphoma
Time to treatment failure | 5 years
  Time to progression
Progression free survival | 5 years
  Duration of survival without relapse or non-relapse mortality
Overall survival | 5 years
  Overall toxicity as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Hawkes, MD, Principal Investigator — Austin Health
Locations (5):
- Australia (5):
  - Ballarat Health, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - St Vincent's Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
IPD is the property of the Sponsor (Austin Health). Results from the research intends to be published/presented in relevant publications/conferences for colleague review

REFERENCES:
- [Derived] Barraclough A, Lee ST, Burgess M, Churilov L, Chong G, Lee D, Gilbertson M, Fancourt T, Manos K, Ritchie DS, Koldej RM, Scott AM, Keane C, Hawkes EA. Nivolumab and rituximab in treatment-naive follicular lymphoma: the phase 2 1st FLOR study. Blood Adv. 2025 Mar 25;9(6):1432-1441. doi: 10.1182/bloodadvances.2024015487. PMID 39853272